CLINICAL TRIAL: NCT05322512
Title: Nectin-4 Targeting ADC Probe for PET Imaging in Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022KT25
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 124I-EV (Experimental): Imaging cohort All enrolled participants will be allocated to undergo three 124I-EV PET/CT scans.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All enrolled participants will be allocated to undergo one 18F-FDG PET/CT scan.

SUMMARY:
To study the normal physiological distribution of the probe 124I-EV in human body and its ability to detect overexpression of Nectin-4 in tumor lesions.

DETAILED DESCRIPTION:
Nectin-4 is highly expressed in different types of cancer and is involved in various aspects of tumor proliferation, angiogenesis, metastasis, tumor recurrence, and DNA repair. Therefore, the development of nuclear medicine molecular probes targeting Nectin-4 is of great significance for improving the specificity and accuracy of Nectin-4 related cancer diagnosis.

EV (Enfortumab vedotin) is the first and only drug targeting Nectin-4 so far. By exploring the diagnostic efficacy of 124I-EV in tumors with high nectin-4 expression, it will not only provide evidence for the early diagnosis of tumors. At the same time, the Nectin-4 expression in tumors can be used to develop effective and precise treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male or female;
2. Patients recommended by clinicians to undergo PET/CT examination for tumor diagnostic staging;
3. The subject patients could fully understand and voluntarily participate in the experiment, and signed the informed consent.
4. Normal heart function;
5. Good follow-up compliance;
6. presence of at least one measurable target lesion according to RECIST1.1 criteria
7. Women of childbearing age (15-49 years) must have a negative pregnancy test within 7 days before the start of the test; Fertile men and women must agree to use effective contraception to prevent pregnancy during the study period and for 3 months after the test.

Exclusion Criteria:

1. Serious abnormality of liver, kidney and blood;
2. Pregnant patients;
3. Pregnant and lactation women;

3) unable to lie flat for half an hour; 4) Refuse to join the clinical investigator; 5) Suffering from claustrophobia or other mental diseases; 6) Other conditions that researchers deem unsuitable for participating in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
SUV (Standardized Uptake Value) | 2 years
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions。 The uptake of the tracer （124I-EV） in tumor lesions by measuring SUV on PET/CT.

IPD SHARING:
Plan to Share IPD: No